CLINICAL TRIAL: NCT04912895
Title: Detection of SARS-CoV-2 RNA and Biomarkers in Coughed Droplets From Patients With COVID-19 and Controls
Brief Title: Detection of SARS-CoV-2 RNA in Coughed Droplets From Patients With COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Georgia Tech Foundation (Other)
Responsible Party: Principal Investigator, Larry J. Anderson, Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00000863
Record Dates: First submitted 2021-06-02; First posted 2021-06-03 (Actual); Results first posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- SARS-CoV-2 Positive (Experimental): Participants who test positive for SARS-CoV-2 with the Polymerase Chain Reaction (PCR) test.
  Interventions: Device: PneumoniaCheck
- Non-COVID-19 Acute Respiratory Illness (Active Comparator): Participants who have an acute respiratory illness other than SARS-CoV-2 infection.
  Interventions: Device: PneumoniaCheck
- Healthy Controls (Other): Participants without any acute respiratory illness.
  Interventions: Device: PneumoniaCheck

INTERVENTIONS:
Device: PneumoniaCheck — Participants are asked to do 5 sets of 10 coughs, with at least 15 minutes between sets, into the PneumoniaCheck device.

SUMMARY:
The purpose of this study is to learn how to better detect infection and understand how severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) causes lung disease and is spread. The novel device called PneumoniaCheck is a safe way to collect material from the lung from coughs. Study participants will collect cough specimens over a 24 hour period.

DETAILED DESCRIPTION:
A novel coronavirus, severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), was detected in association with cases of severe respiratory illness and pneumonia (COVID-19) in Wuhan City, Hubei Province, China in December 2019. The virus subsequently spread widely throughout China and globally. Addressing this unprecedented global pandemic is requiring all available tools to diagnose infection, manage ill patients, understand disease pathogenesis and virus transmission to guide efforts to decrease transmission and rapidly develop anti-viral drugs and vaccines. The researchers of this study propose to use the PneumoniaCheck™, a device developed collaboratively by investigators at the Georgia Institute of Technology (GA Tech) and the Centers for Disease Control and Prevention (CDC), to help address these issues. This device, non-invasively, captures coughed droplets onto a filter with minimal contamination from upper airway secretions. In preliminary studies in cystic fibrosis, mycobacterium tuberculosis (TB) patients and control patients, the researchers detected bacterial DNA by PCR, inflammatory cytokines and chemokines by multiplex Luminex assays, surfactant by enzyme immunoassay (EIA), and amylase by enzymatic assay. These data show that this device can provide high quality specimens from the lung with minimal risk to the patient and healthcare provider and much lower risk than invasive procedures such as bronchioloalveolar lavage. In addition, with this device, the researchers can acquire specimens from patients who do not have a productive cough (dry cough), a commonly reported symptom for COVID-19, and specimens with minimal upper respiratory contamination unlike a sputum specimen. Thus, this device can provide lung secretion specimens to improve detection of SARS-CoV-2 RNA (lung specimens are better for detecting virus than upper respiratory tract specimens) and detect inflammatory and other biomarkers to explore pathogenesis of disease, identify inflammatory processes that might be amenable to intervention, and identify biomarkers of disease severity for patient management and evaluation of vaccines and anti-viral drugs. The goal of this study is to determine how PneumoniaCheck™ can help diagnose, manage, and understand pathogenesis of disease and transmission risk of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Being treated for an acute respiratory illness either as inpatients or outpatients at Emory University Hospital
* English is a primary spoken language

Exclusion Criteria:

* none

Inclusion Criteria for Healthy Volunteers:

* Prior registration in an adult participant database and agreed to be contacted for future studies
* English is a primary spoken language

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry Anderson, MD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory Children's Center, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Wesley Woods Center, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data collected during the trial will be made available for sharing, after deidentification, as consistent with Health Information Privacy and Portability Act (HIPPA) regulations.
Supporting Information: Study Protocol
Time Frame: Data will be available for sharing following the publication of manuscripts related to the primary aims of this study.
Access Criteria: Individual participant data will be available for sharing with researchers who provide a methodologically sound proposal, in order to achieve the aims stated in the approved proposal. Proposals should be directed to Dr. Larry Anderson.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Emory Children's Center, Emory University Hospital Midtown, Emory University Hospital, and the Wesley Woods Center in Atlanta, Georgia, USA. Participant enrollment began April 14, 2022 and all follow-up assessments were completed by August 5, 2022.
Pre-assignment Details: The study initially planned to recruit participants with non-coronavirus disease 2019 (COVID-19) respiratory illness, however, resources did not permit including this study arm.
Groups:
- PneumoniaCheck Among SARS-CoV-2 Positive Participants: Participants who test positive for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) with the polymerase chain reaction (PCR) test use the PneumoniaCheck device to collect material from the lung from coughs. Participants are asked to do 5 sets of 10 coughs, with at least 15 minutes between sets, into the PneumoniaCheck device.
- PneumoniaCheck Among Non-COVID-19 Acute Respiratory IllnessParticipants: Participants who have an acute respiratory illness other than SARS-CoV-2 infection use the PneumoniaCheck device to collect material from the lung from coughs. Participants are asked to do 5 sets of 10 coughs, with at least 15 minutes between sets, into the PneumoniaCheck device.
- PneumoniaCheck Among Healthy Controls: Participants without any acute respiratory illness use the PneumoniaCheck device to collect material from the lung from coughs. Participants are asked to do 5 sets of 10 coughs, with at least 15 minutes between sets, into the PneumoniaCheck device.
Period: Overall Study
Arm/Group | PneumoniaCheck Among SARS-CoV-2 Positive Participants | PneumoniaCheck Among Non-COVID-19 Acute Respiratory IllnessParticipants | PneumoniaCheck Among Healthy Controls
Started | 51 | 0 | 18
Completed | 49 | 0 | 18
Not Completed | 2 | 0 | 0
Not completed — Unable to provide specimen | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- PneumoniaCheck Among SARSCoV-2 Positive Participants: Participants who test positive for SARS-CoV-2 with the PCR test use the PneumoniaCheck device to collect material from the lung from coughs. Participants are asked to do 5 sets of 10 coughs, with at least 15 minutes between sets, into the PneumoniaCheck device.
- Total: Total of all reporting groups
Arm/Group | PneumoniaCheck Among SARSCoV-2 Positive Participants | PneumoniaCheck Among Healthy Controls | Total
Number analyzed (Participants) | 51 | 18 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 18 | 69
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 27 | 0 | 27
  Male | 21 | 0 | 21
  Not collected | 3 | 18 | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 51 | 18 | 69

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of Detecting SARS-CoV-2 RNA
Description: The number of correct identification of participants with SARS-CoV-2 infection (true positives) detected by RNA in cough-generated droplets captured with the PneumoniaCheck.
Time Frame: Up to Hour 24
Population: This analysis includes participants who successfully provided a cough sample using the PneumoniaCheck.
Measure: Count of Participants; unit: Participants
Arm/Group | PneumoniaCheck Among SARSCoV-2 Positive Participants | PneumoniaCheck Among Healthy Controls
Number analyzed (Participants) | 49 | 18
Participants | 31 | 0

2. Primary Outcome: Specificity of Detecting SARS-CoV-2 RNA
Description: The number of correct identification of participants without SARS-CoV-2 infection (true negatives) detected by RNA in cough-generated droplets captured with the PneumoniaCheck.
Time Frame: Up to Hour 24
Population: This analysis includes participants who successfully provided a cough sample using the PneumoniaCheck.
Measure: Count of Participants; unit: Participants
Arm/Group | PneumoniaCheck Among SARSCoV-2 Positive Participants | PneumoniaCheck Among Healthy Controls
Number analyzed (Participants) | 49 | 18
Participants | 10 | 18

3. Other Pre Specified Outcome: Amount of IFN Gamma Detected
Description: The researchers detected biomarkers of inflammation in coughed specimens from patient with COVID-19 hypothesizing that biomarkers of inflammation from the lung will indicate disease activity, informing pathogenesis of COVID-19 disease. The value of detecting inflammatory cytokines, including IFN gamma, in cough-generated droplets with PneumoniaCheck from COVID-19 patients will be evaluated.
Time Frame: Up to Hour 24
Population: This analysis includes participants who successfully provided a cough sample using the PneumoniaCheck.
Measure: Median (Full Range); unit: picograms per milliliter (pg/mL)
Arm/Group | PneumoniaCheck Among SARSCoV-2 Positive Participants | PneumoniaCheck Among Healthy Controls
Number analyzed (Participants) | 49 | 18
picograms per milliliter (pg/mL) | 0.201 [0.029 to 0.342] | 0.229 [0.003 to 2.222]

4. Other Pre Specified Outcome: Amount of Interleukin (IL)-1 Beta Detected
Description: The researchers detected biomarkers of inflammation in coughed specimens from patient with COVID-19 hypothesizing that biomarkers of inflammation from the lung will indicate disease activity, informing pathogenesis of COVID-19 disease. The value of detecting inflammatory cytokines, including IL-1 beta, in cough-generated droplets with PneumoniaCheck from COVID-19 patients will be evaluated.
Time Frame: Up to Hour 24
Population: This analysis includes participants who successfully provided a cough sample using the PneumoniaCheck.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | PneumoniaCheck Among SARSCoV-2 Positive Participants | PneumoniaCheck Among Healthy Controls
Number analyzed (Participants) | 49 | 18
pg/mL | 0.140 [0.052 to 0.566] | 0.131 [0.076 to 64.522]

5. Other Pre Specified Outcome: Amount of IL-2 Detected
Description: as for outcome 4
Time Frame: Up to Hour 24
Population: This analysis includes participants who successfully provided a cough sample using the PneumoniaCheck.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | PneumoniaCheck Among SARSCoV-2 Positive Participants | PneumoniaCheck Among Healthy Controls
Number analyzed (Participants) | 49 | 18
pg/mL | 0.157 [0.071 to 0.271] | 0.219 [0.117 to 1.355]

6. Other Pre Specified Outcome: Amount of IL-4 Detected
Description: The researchers detected biomarkers of inflammation in coughed specimens from patient with COVID-19 hypothesizing that biomarkers of inflammation from the lung will indicate disease activity, informing pathogenesis of COVID-19 disease. The value of detecting inflammatory cytokines, including IL-4, in cough-generated droplets with PneumoniaCheck from COVID-19 patients will be evaluated.
Time Frame: Up to Hour 24
Population: This analysis includes participants who successfully provided a cough sample using the PneumoniaCheck.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | PneumoniaCheck Among SARSCoV-2 Positive Participants | PneumoniaCheck Among Healthy Controls
Number analyzed (Participants) | 49 | 18
pg/mL | 0.009 [0.004 to 0.041] | 0.009 [0.003 to 0.104]

7. Other Pre Specified Outcome: Amount of IL-6 Detected
Description: The researchers detected biomarkers of inflammation in coughed specimens from patient with COVID-19 hypothesizing that biomarkers of inflammation from the lung will indicate disease activity, informing pathogenesis of COVID-19 disease. The value of detecting inflammatory cytokines, including IL-6, in cough-generated droplets with PneumoniaCheck from COVID-19 patients will be evaluated.
Time Frame: Up to Hour 24
Population: This analysis includes participants who successfully provided a cough sample using the PneumoniaCheck.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | PneumoniaCheck Among SARSCoV-2 Positive Participants | PneumoniaCheck Among Healthy Controls
Number analyzed (Participants) | 49 | 18
pg/mL | 0.081 [0.020 to 0.531] | 0.076 [0.001 to 3.763]

8. Other Pre Specified Outcome: Amount of IL-8 Detected
Description: The researchers will detect biomarkers of inflammation in coughed specimens from patient with COVID-19 hypothesizing that biomarkers of inflammation from the lung will indicate disease activity, informing pathogenesis of COVID-19 disease. The value of detecting inflammatory cytokines, including IL-8, in cough-generated droplets with PneumoniaCheck from COVID-19 patients will be evaluated.
Time Frame: Up to Hour 24
Population: This analysis includes participants who successfully provided a cough sample using the PneumoniaCheck.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | PneumoniaCheck Among SARSCoV-2 Positive Participants | PneumoniaCheck Among Healthy Controls
Number analyzed (Participants) | 49 | 18
pg/mL | 0.132 [0.037 to 9.984] | 0.095 [0.019 to 639.432]

9. Other Pre Specified Outcome: Amount of IL-10 Detected
Description: The researchers detected biomarkers of inflammation in coughed specimens from patient with COVID-19 hypothesizing that biomarkers of inflammation from the lung will indicate disease activity, informing pathogenesis of COVID-19 disease. The value of detecting inflammatory cytokines, including IL-10, in cough-generated droplets with PneumoniaCheck from COVID-19 patients will be evaluated.
Time Frame: Up to Hour 24
Population: This analysis includes participants who successfully provided a cough sample using the PneumoniaCheck.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | PneumoniaCheck Among SARSCoV-2 Positive Participants | PneumoniaCheck Among Healthy Controls
Number analyzed (Participants) | 49 | 18
pg/mL | 0.028 [0.015 to 0.113] | 0.031 [0.019 to 0.634]

10. Other Pre Specified Outcome: Amount of IL-12p70 Detected
Description: The researchers detected biomarkers of inflammation in coughed specimens from patient with COVID-19 hypothesizing that biomarkers of inflammation from the lung will indicate disease activity, informing pathogenesis of COVID-19 disease. The value of detecting inflammatory cytokines, including IL-12p70, in cough-generated droplets with PneumoniaCheck from COVID-19 patients will be evaluated.
Time Frame: Up to Hour 24
Population: This analysis includes participants who successfully provided a cough sample using the PneumoniaCheck.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | PneumoniaCheck Among SARSCoV-2 Positive Participants | PneumoniaCheck Among Healthy Controls
Number analyzed (Participants) | 49 | 18
pg/mL | 0.088 [0.040 to 0.130] | 0.082 [0.033 to 0.543]

11. Other Pre Specified Outcome: Amount of IL-13 Detected
Description: The researchers detected biomarkers of inflammation in coughed specimens from patient with COVID-19 hypothesizing that biomarkers of inflammation from the lung will indicate disease activity, informing pathogenesis of COVID-19 disease. The value of detecting inflammatory cytokines, including IL-13, in cough-generated droplets with PneumoniaCheck from COVID-19 patients will be evaluated.
Time Frame: Up to Hour 24
Population: This analysis includes participants who successfully provided a cough sample using the PneumoniaCheck.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | PneumoniaCheck Among SARSCoV-2 Positive Participants | PneumoniaCheck Among Healthy Controls
Number analyzed (Participants) | 49 | 18
pg/mL | 0.618 [0.364 to 0.708] | 0.420 [0.141 to 7.549]

12. Other Pre Specified Outcome: Amount of Tumour Necrosis Factor (TNF) Alpha Detected
Description: The researchers detected biomarkers of inflammation in coughed specimens from patient with COVID-19 hypothesizing that biomarkers of inflammation from the lung will indicate disease activity, informing pathogenesis of COVID-19 disease. The value of detecting inflammatory cytokines, including TNF alpha, in cough-generated droplets with PneumoniaCheck from COVID-19 patients will be evaluated.
Time Frame: Up to Hour 24
Population: This analysis includes participants who successfully provided a cough sample using the PneumoniaCheck.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | PneumoniaCheck Among SARSCoV-2 Positive Participants | PneumoniaCheck Among Healthy Controls
Number analyzed (Participants) | 49 | 18
pg/mL | 0.026 [0.004 to 0.086] | 0.017 [0.001 to 2.211]

13. Other Pre Specified Outcome: Detection of Interleukin (IL)-1 Alpha
Description: The researchers will detect biomarkers of inflammation in coughed specimens from patient with COVID-19 hypothesizing that biomarkers of inflammation from the lung will indicate disease activity, informing pathogenesis of COVID-19 disease. The value of detecting inflammatory cytokines, including IL-1 alpha, in cough-generated droplets with PneumoniaCheck from COVID-19 patients will be evaluated.
Time Frame: Up to Hour 24
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Detection of Interferon (IFN) Alpha
Description: The researchers will detect biomarkers of inflammation in coughed specimens from patient with COVID-19 hypothesizing that biomarkers of inflammation from the lung will indicate disease activity, informing pathogenesis of COVID-19 disease. The value of detecting inflammatory cytokines, including IFN alpha, in cough-generated droplets with PneumoniaCheck from COVID-19 patients will be evaluated.
Time Frame: Up to Hour 24
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Detection of Granulocyte-macrophage Colony-stimulating Factor (GM-CSF)
Description: The researchers will detect biomarkers of inflammation in coughed specimens from patient with COVID-19 hypothesizing that biomarkers of inflammation from the lung will indicate disease activity, informing pathogenesis of COVID-19 disease. The value of detecting inflammatory cytokines, including GM-CSF, in cough-generated droplets with PneumoniaCheck from COVID-19 patients will be evaluated.
Time Frame: Up to Hour 24
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Detection of IL-17A
Description: The researchers will detect biomarkers of inflammation in coughed specimens from patient with COVID-19 hypothesizing that biomarkers of inflammation from the lung will indicate disease activity, informing pathogenesis of COVID-19 disease. The value of detecting inflammatory cytokines, including IL-17A, in cough-generated droplets with PneumoniaCheck from COVID-19 patients will be evaluated.
Time Frame: Up to Hour 24
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Detection of Interferon Gamma-induced Protein 10 (IP-10) C-X-C Motif Chemokine Ligand 10 (CXCL10)
Description: The researchers will detect biomarkers of inflammation in coughed specimens from patient with COVID-19 hypothesizing that biomarkers of inflammation from the lung will indicate disease activity, informing pathogenesis of COVID-19 disease. The value of detecting inflammatory chemokines, including IP-10, also known as C-X-C motif chemokine ligand 10 (CXCL10), in cough-generated droplets with PneumoniaCheck from COVID-19 patients will be evaluated.
Time Frame: Up to Hour 24
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Detection of Macrophage Inflammatory Protein-1 (MIP-1) Alpha
Description: The researchers will detect biomarkers of inflammation in coughed specimens from patient with COVID-19 hypothesizing that biomarkers of inflammation from the lung will indicate disease activity, informing pathogenesis of COVID-19 disease. The value of detecting inflammatory chemokines, including MIP-1 alpha, also known as C-C motif chemokine ligand 3 (CCL3), in cough-generated droplets with PneumoniaCheck from COVID-19 patients will be evaluated.
Time Frame: Up to Hour 24
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Detection of Monocyte Chemoattractant Protein 1 (MCP-1)
Description: The researchers will detect biomarkers of inflammation in coughed specimens from patient with COVID-19 hypothesizing that biomarkers of inflammation from the lung will indicate disease activity, informing pathogenesis of COVID-19 disease. The value of detecting inflammatory chemokines, including MCP-1, also known as C-C motif chemokine ligand 2 (CCL2), in cough-generated droplets with PneumoniaCheck from COVID-19 patients will be evaluated.
Time Frame: Up to Hour 24
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Detection of Surfactant A
Description: The researchers will detect biomarkers of inflammation in coughed specimens from patient with COVID-19 hypothesizing that biomarkers of inflammation from the lung will indicate disease activity, informing pathogenesis of COVID-19 disease. The value of detecting surfactant A chemokines in cough-generated droplets with PneumoniaCheck from COVID-19 patients will be evaluated.
Time Frame: Up to Hour 24
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Detection of MIP-1 Beta
Description: The researchers will detect biomarkers of inflammation in coughed specimens from patient with COVID-19 hypothesizing that biomarkers of inflammation from the lung will indicate disease activity, informing pathogenesis of COVID-19 disease. The value of detecting inflammatory chemokines, including MIP-1 beta, also known as C-C motif chemokine ligand 4 (CCL4), in cough-generated droplets with PneumoniaCheck from COVID-19 patients will be evaluated.
Time Frame: Up to Hour 24
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected during the time period of specimen collection, up to 24 hours.
Description: Only adverse events occurring during specimen collection were collected.
Arm/Group | PneumoniaCheck Among SARSCoV-2 Positive Participants | PneumoniaCheck Among Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/18
Other Adverse Events (participants affected / at risk) | 0/51 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2021-09-10): https://cdn.clinicaltrials.gov/large-docs/95/NCT04912895/Prot_001.pdf